CLINICAL TRIAL: NCT00257140
Title: A Multicenter, Active-Controlled, Randomized Study to Evaluate the Safety and Efficacy of Oral Levofloxacin Versus Cefaclor in the Treatment of Acute Bacterial Exacerbation of Chronic Bronchitis in Adults
Brief Title: A Study of the Safety and Effectiveness of Levofloxacin Compared With Cefaclor in the Treatment of Adults With Chronic Bronchitis Experiencing Rapid Onset of Worsening of Symptoms Caused by Bacteria
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005494
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-01

CONDITIONS: Bronchitis; Bronchitis, Chronic
Keywords: Bronchitis; chronic bronchitis; lung diseases; respiratory tract infections; bronchial diseases; antibacterial agents; quinolones; levofloxacin
MeSH Terms: conditions — Bronchitis; Bronchitis, Chronic; Lung Diseases; Respiratory Tract Infections; Bronchial Diseases | interventions — Levofloxacin

INTERVENTIONS:
Drug: levofloxacin

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of levofloxacin, an antibiotic, compared with cefaclor, another antibiotic, in the treatment of adults with chronic bronchitis experiencing rapid onset of worsening of symptoms caused by bacteria.

DETAILED DESCRIPTION:
This is a randomized, open-label, parallel group, multicenter study to determine the effectiveness and safety of 488 mg of levofloxacin (once daily by mouth for 5 - 7 days) compared with 250 mg of cefaclor (every 8 hours for 7 - 10 days) in adults with chronic bronchitis experiencing rapid onset of worsening of symptoms caused by bacterial infection. The study consists of 3 visits: one visit for screening and enrollment, and 2 visits for assessment of safety and effectiveness (one visit on Days 3 - 5 of the study and one visit [post-therapy] 5 - 7 days after the last dose of the study drug). The total duration of patient participation in the study is approximately 2 weeks. Levofloxacin and cefaclor are antibacterial agents used for the treatment of many types of infections, including infections with a rapid onset and brief duration caused by bacteria. The primary assessment of effectiveness in this study is the microbiologic response to treatment (the rate of elimination of disease-causing bacteria, by patient, and by type of bacteria), 5 - 7 days after the last dose of study drug. Safety evaluations (incidence of adverse events, physical examination, laboratory tests) are performed throughout the study. The study hypothesis is that treatment with levofloxacin is at least as effective and as well tolerated as treatment with cefaclor in adult patients with chronic bronchitis experiencing sudden worsening of symptoms caused by bacterial infection. Levofloxacin 488 mg by mouth once daily for 5 - 7 days, or cefaclor 250 mg by mouth every 8 hours for 7 - 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic bronchitis with a rapid onset of worsening of symptoms caused by bacteria
* history of chronic obstructive lung disease (chronic bronchitis and/or emphysema)
* recent increase in cough
* change in type of sputum (the mucus produced on coughing) and/or an increase in the production of sputum
* received previous antibiotic treatment if the previous treatment lasted for 24 hours or less, or if the previous treatment lasted longer than 24 hours but there was no improvement or stabilization of the disease.

Exclusion Criteria:

* Illness requiring antibiotic treatment by injection into a vein, beneath the skin, or into a muscle, or has a requirement of an antibiotic medication taken orally in addition to the study drug
* infection due to bacteria known (prior to the start of the study) to be resistant to the study drug
* previous allergic or serious adverse reaction to similar antibiotics
* diagnosis of pneumonia, determined by a chest x-ray at the start of the trial
* has cystic fibrosis, seizure disorders, kidney disease, or an unstable psychiatric condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 1931-06; Study Completion 1994-07 (Actual)

PRIMARY OUTCOMES:
Rate of elimination of disease-causing bacteria, by patient, and by type of bacteria, 5 - 7 days after the last dose of study drug.

SECONDARY OUTCOMES:
Clinical response rate (reduction in signs and symptoms) at post-therapy (5 - 7 days after the last dose of study drug). Incidence of adverse events; changes in physical examination and laboratory tests after treatment with the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Habib MP, Gentry LO, et al. Multicenter, randomized study comparing efficacy and safety of oral levofloxacin and cefaclor in treatment of acute bacterial exacerbations of chronic bronchitis, Infectious Diseases in Clinical Practice 1998;7:101-109
- See also: A study of the safety and effectiveness of levofloxacin compared to cefaclor in the treatment of adults with chronic bronchitis experiencing rapid onset of worsening of symptoms caused by bacteria — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=657&filename=CR005494_CSR.pdf